CLINICAL TRIAL: NCT06192901
Title: A Limited Patient Cohort Follow-up Study to Assess the Long-term Safety and Performance of Hydrophobic and Hydrophilic Intraocular Lenses in Bilateral Cataract Surgery
Brief Title: Safety and Performance of Hydrophobic and Hydrophilic Intraocular Lenses After Bilateral Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AT ELANA 841P-BER-401-23
Record Dates: First submitted 2023-09-12; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-09

CONDITIONS: Senile Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study eye AT ELANA 841P: Subjects who underwent bilateral cataract surgery with the implantation of the IOL AT ELANA 841P in the first eye.
- Study eye AT LISA 839MP: Subjects who underwent bilateral cataract surgery with the implantation of the IOL AT LISA tri 839MP in the second eye.

SUMMARY:
Subjects who had a bilateral age-related cataract surgery with the IOLs AT ELANA 841P and AT LISA tri 839MP will be contacted and invited to attend a postoperative visit more than one year after the surgery

DETAILED DESCRIPTION:
The main objective of this clinical investigation is to collect data on the IOLs AT ELANA 841P and AT LISA tri 839MP in subjects who underwent bilateral cataract surgery with the use of the two different types of IOLs to confirm the long-term performance and safety of the IOLs.

Retro-prospective, comparative, non-interventional, non-randomized, single center study on medical devices with one follow-up visit after more than 12 months of a bilateral cataract surgery.Subjects who had a bilateral age-related cataract surgery with the IOLs AT ELANA 841P and AT LISA tri 839MP will be contacted and invited to attend a postoperative visit more than one year after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient of any gender;
2. Patients who had an uncomplicated (no intra-operative complication) age-related cataract surgery
3. Currently implanted with an IOL model AT ELANA 841P into the capsular bag in one eye and with the IOL model AT LISA tri 839MP into the capsular bag of the other eye.
4. The postoperative visit was scheduled to be conducted more than one year after the second eye surgery.
5. Given written informed consent by patient.

Exclusion Criteria:

1. Patients unable to meet the limitations of the protocol or likely of non-cooperation during the study
2. Patient whose freedom is impaired by administrative or legal order
3. Concurrent participation in another drug or device investigation that could confound the outcome of this investigation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to 20 eyes in 10 adult subjects who underwent bilateral cataract surgery with the implantation of the IOL AT ELANA 841P in the first eye and AT LISA tri 839MP in the second eye.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Monocular Corrected Distance Visual Acuity (CDVA) | 12 to 24 months after cataract surgery
Slit Lamp Examination | 12 to 24 months after cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Quesada, San Salvador, El Salvador